CLINICAL TRIAL: NCT06461871
Title: Combined Effects of Balance Training With Moderate Intensity Aerobic Versus Resisted Training on Glycemic Control, Cardiorespiratory Fitness , and Quality of Life in Patients With Type 2 Diabetes Milletus.
Brief Title: Combined Effects of BT With Moderate Intensity Aerobic Versus RT in Type 2 DM.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0337
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cardio respiratory fitness; aerobic exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Group A received moderate intensity aerobic exercises which include walking, cycling, with each session lasting 15 minutes for 3-5 days per week in combination with balance training which include heel raise, standing march with 10 repetitions each for 3-5 days per week. Group B receive moderate intensity resistance exercises which include biceps curls, triceps curls , with each session lasting 10 repetitions for 3-5 days per week in combination with balance training which include heel raise, standing march with 10 repetitions each for 3-5 days per week. The study will be completed with time duration of six months .Primary outcome of research will be glycemic control, cardio respiratory fitness, and quality of life.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate intensity aerobic exercises with balance training (Experimental): A received moderate intensity aerobic exercises which include walking, cycling, with each session lasting 15 minutes for 3-5 days per week in combination with balance training which include heel raise
  Interventions: Other: BALANCE TRAINING WITH MODERATE INTESITY AEROBIC VERSUS RESISTED TRAINING (RT); Other: Moderate intensity resistance exercises in combination with balance training
- moderate intensity resistance exercises with balance training (Experimental): Group B receive moderate intensity resistance exercises which include biceps curls, triceps curls , with each session lasting 10 repetitions for 3-5 days per week in combination with balance training which include heel raise
  Interventions: Other: BALANCE TRAINING WITH MODERATE INTESITY AEROBIC VERSUS RESISTED TRAINING (RT); Other: Moderate intensity resistance exercises in combination with balance training

INTERVENTIONS:
Other: BALANCE TRAINING WITH MODERATE INTESITY AEROBIC VERSUS RESISTED TRAINING (RT) — The duration of study is 6 months. Three to five sessions of both aerobic and resistance exercise training in combination with balance training are taken out per week . Each session lasting 15 minutes. GROUP A: Baseline treatment + Moderate intensity aerobic exercises in combination with balance training
  Other Names: Moderate intensity aerobic exercises in combination with balance training
Other: Moderate intensity resistance exercises in combination with balance training — The duration of study is 6 months. Three to five sessions of both aerobic and resistance exercise training in combination with balance training are taken out per week . Each session lasting 15 minutes. GROUP B: Baseline treatment + Moderate intensity resistance exercises in combination with balance training

SUMMARY:
A randomized control trail will be conducted at Social Security Teaching Hospital, Multan Road, Lahore. Social Security Teaching Hospital Shah rah, Lahore. Non -probability Convenient Random Sampling Technique will be applied on patients who will be allocated through simple random sampling into group A and group B. Group A received moderate intensity aerobic exercises which include walking, cycling, with each session lasting 15 minutes for 3-5 days per week in combination with balance training which include heel raise, standing march with 10 repetitions each for 3-5 days per week. Group B receive moderate intensity resistance exercises which include biceps curls, triceps curls , with each session lasting 10 repetitions for 3-5 days per week in combination with balance training which include heel raise, standing march with 10 repetitions each for 3-5 days per week. The study will be completed with time duration of six months .Primary outcome of research will be glycemic control, cardio respiratory fitness, and quality of life. Data will be analyzed using SPSS software version 21. After assessing normality of Shapiro-will test, it will be decided either parametric or non parametric test will be used within a group or between groups.

DETAILED DESCRIPTION:
Exercise is often authorize for type 2 diabetic patients in command to intensify their physical activity, physical fitness, and glycolic management . More than 95 of individuals with diabetes have type 2 diabetes millets (DM), which is initiated by body inappropriate utilization of insulin .Type 2 diabetes has been associated to sedentary habits, smoking, immoderate alcohol use, extreme glucose intake, among other lifestyle representative. Diabetic neuropathy is frequent complication of type 2 diabetes millets with a considerable effect on health of influenced individuals .The existence of diabetic neuropathy may impair balance in affected patients. Type 2 diabetes millets can remarkably lesser person's quality of life, with health related quality of life constitute the main concern.

A randomized control trail will be conducted at Social Security Teaching Hospital, Multan Road, Lahore. Social Security Teaching Hospital Shah rah, Lahore. Non -probability Convenient Random Sampling Technique will be applied on patients who will be allocated through simple random sampling into group A and group B. Group A received moderate intensity aerobic exercises which include walking, cycling, with each session lasting 15 minutes for 3-5 days per week in combination with balance training (BT) which include heel raise, standing march with 10 repetitions each for 3-5 days per week. Group B receive moderate intensity resistance exercises which include biceps curls, triceps curls , with each session lasting 10 repetitions for 3-5 days per week in combination with balance training which include heel raise, standing march with 10 repetitions each for 3-5 days per week. The study will be completed with time duration of six months .Primary outcome of research will be glycemic control, cardio respiratory fitness, and quality of life. Data will be analyzed using SPSS software version 21. After assessing normality of Shapiro-will test, it will be decided either parametric or non parametric test will be used within a group or between groups.

Key words:

Type 2 diabetes millets, cardio respiratory fitness, glycemic control, aerobic exercise, resisted exercise,

ELIGIBILITY:
Inclusion Criteria:

* Participants with 40-60 years of age with type 2 diabetes mellitus.(16)
* Both male and female participants are included in study.(17)
* Participants with HbA1c level greater than >6.4(18)
* Patients with diabetic neuropathy (19)
* Without participation in any supervised exercise program in last 6 months(19, 20)
* Dietary pattern stabilized for at least 6 months(8)

Exclusion Criteria:

* Participants with mental impairments .(21, 22)
* Those with gout or hyperuricemia. (16, 22, 23)
* Patient with serious cardiovascular risk factors (24, 25)
* Pregnant females (26, 27)
* Participants with hepatic and renal impairment.(22)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
VO2 MAX | 12 weeks
  To assess cardiorespiratory fitness , also known as maximal oxygen uptake , measures maximum amount of oxygen a person can utilize oxygen.
  VO2 max = 132.853 - (0.0769 x your weight in pounds) - (0.3877 x your age) + (6.315 if you are male or 0 if you are female) - (3.2649 x your walking time) - (0.1565 x your heart rate at the end of the test).
EQ -5D-5L QUESTIONNAIRE | 12 weeks
  EQ-5D-5L is a self assessed , health related, quality of life questionnaire. The scale measures quality of life on a 5 component scale including mobility, self care, usual activities, pain/discomfort , anxiety /depression .
HbA1c | 12 weeks
  Hemoglobin analyzers (also referred to as HbA1c Analyzer) can report the concentration of hemoglobin in a blood or urine sample in g/L, g/dL, or mol/L. HbA1c Analyzers can run tests with samples as small as 1uL in just a few minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Study Chair — Riphah International University
Locations (1):
- Social Security Teaching Hospital Shah rah, Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawite F, Girma M, Shibiru T, Kefelew E, Hailu T, Temesgen R, Abebe G. Factors associated with poor glycemic control among adult patients with type 2 diabetes mellitus in Gamo and Gofa zone public hospitals, Southern Ethiopia: A case-control study. PLoS One. 2023 Mar 10;18(3):e0276678. doi: 10.1371/journal.pone.0276678. eCollection 2023. PMID 36897872
- [Background] Lim JU, Park CK, Kim TH, Jang AS, Park YB, Rhee CK, Jung KS, Yoo KH, Lee WY, Yoon HK. The Difficulty Of Improving Quality Of Life In COPD Patients With Depression And Associated Factors. Int J Chron Obstruct Pulmon Dis. 2019 Oct 9;14:2331-2341. doi: 10.2147/COPD.S216746. eCollection 2019. PMID 31632002